CLINICAL TRIAL: NCT04731844
Title: Efficacy of Curcumin and Piperine in Patients on Active Surveillance for Either Monoclonal Gammopathy of Unknown Significance (MGUS), Low-risk Smoldering Multiple Myeloma (SMM) or Early Stage Prostate Cancer: A Pilot Study
Brief Title: Curcumin and Piperine in Patients on Surveillance for Monoclonal Gammopathy, Smoldering Myeloma or Prostate Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Brea Lipe, Professor - Department of Medicine , Hematology/Oncology (SMD), University of Rochester
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMLT20123
Record Dates: First submitted 2021-01-26; First posted 2021-02-01 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Prostate Cancer; Multiple Myeloma; Smoldering Multiple Myeloma (SMM); Monoclonal Gammopathy of Undetermined Significance
Keywords: curcumin; peperine; prostate cancer; Multiple Myeloma; Smoldering Multiple Myeloma (SMM); Monoclonal Gammopathy of Undetermined Significance (MGUS)
MeSH Terms: conditions — Prostatic Neoplasms; Multiple Myeloma; Smoldering Multiple Myeloma; Monoclonal Gammopathy of Undetermined Significance | interventions — Curcumin; piperine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Prostate Cancer (Experimental): Curcumin plus Piperine at a dose of 4 gram/5mg orally BID for 12 months
  Interventions: Drug: Curcumin plus Piperine
- Smoldering Multiple Myeloma (SMM) (Experimental): Curcumin plus Piperine at a dose of 4 gram/5mg orally BID for 12 months
  Interventions: Drug: Curcumin plus Piperine
- Monoclonal Gammopathy of Unknown Significance (MGUS) (Experimental): Curcumin plus Piperine at a dose of 4 gram/5mg orally BID for 12 months
  Interventions: Drug: Curcumin plus Piperine

INTERVENTIONS:
Drug: Curcumin plus Piperine — Curcumin with piperine is a well-tolerated over-the-counter supplement.
  Other Names: Curcumin C3 Complex®

SUMMARY:
To explore the use of curcumin and piperine supplementation at a dose of 4 gram/5mg twice a day in early stage prostate cancer patient undergoing active surveillance or patients on observation for MGUS/ low-risk smoldering myeloma.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether the supplement of curcumin plus peperine can prevent or delay the progression of prostate cancer, monoclonal gammopathy of unknown significant, or low-risk smoldering myeloma into a more aggressive cancer which requires treatment. The investigator will be evaluating a marker in patients blood called MIC-1 to determine whether it could be a useful predictor of whether the disease is improving or progressing.

ELIGIBILITY:
Inclusion Criteria:

* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry.
* Age ≥ 18 years of age.
* Karnofsky performance status (KPS) of ≥ 70%.
* Subjects with either 1) non-metastatic biopsy proven adenocarcinoma of the prostate who have chosen AS the treatment option for their prostate cancer or 2) have the diagnosis of either MGUS or low-risk SMM and are currently on observation alone.
* For patients with MGUS or low-risk SMM, diagnosis must be according to the definition of the International Myeloma Working Group (IMWG).

  1. MGUS: serum M-protein <3.0g/dL, <10% clonal plasma cells (PCs) in the bone marrow, and absence of end-organ damage (CRAB criteria) that can be attributed to the plasma cell disorder.
  2. SMM: serum M-protein of ≥3.0g/dL or a proportion of clonal PCs in the BM of ≥10% but <60%, and no evidence of end organ damage as described below.

     * Absence of end organ damage is defined by absence of CRAB criteria:

       * C: Absence of hypercalcemia, defined as calcium ≤11mg/dL.
       * R: Absence of renal failure, defined as serum creatinine ≤2.0mg/dL.
       * A: Absence of anemia, defined as hemoglobin ≥10g/dL.
       * B: Absence of lytic bone lesions per IMWG recommendations: One of either PET-CT, low-dose whole-body CT, or whole- body MRI. Increased uptake on PET-CT alone is not adequate for the diagnosis of multiple myeloma; evidence of underlying osteolytic bone destruction is needed on the CT portion of the examination.
* At least one of the risk factors below that portends for an increased risk of progression to MM:

  * Abnormal serum free light chain ratio.
  * M-spike ≥2.0g/dL.
  * ≥ 20% bone marrow clonal plasma cells.
  * Immunoparesis ≥20% reduction from institutional normal standard of uninvolved immunoglobulins.

Exclusion Criteria

* Currently taking supplements containing either curcumin or piperine.
* Plan to start any additional over the counter supplements prior to or during trial period.
* For prostate cancer patients must not be planning to undergoing primary curative therapy for their prostate cancer (radiation, surgery, brachytherapy).
* For MGUS/ SMM patients, must not have had evidence of disease progression which might require treatment during the one-year study period.
* Other: symptomatic plasma cell leukemia, amyloidosis, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein).
* Subject is pregnant or breast feeding, or planning to become pregnant during the treatment period.
* Evidence of any of the following conditions per subject self-report or medical chart review: Major surgery or significant traumatic injury occurring within 4 weeks before enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-12-14 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Response rate of Curcumin & Piperine supplementation in patients on AS for either early stage prostate cancer or MGUS. | From date of enrollment until the date of first documented response assessed up to 12 months
  Measure of time from study enrollment until response

SECONDARY OUTCOMES:
Progression Free Survival | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  Measure of time from study enrollment until progression.

CONTACTS AND LOCATIONS:
Overall Officials: Brea Lipe, Principal Investigator — University of Rochester Wilmot Cancer Center
Locations (1):
- University of Rochester, Rochester, New York, United States